CLINICAL TRIAL: NCT06519500
Title: Generation of Organoids of Neuroendocrine Neoplasms of the Gastro-Entero-Pancreatic Tract Obtained From Patients Undergoing Surgery
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1823/23
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Gastro-entero-pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgery for neuroendocrine neoplasia: At least 10 cultures of organoids of Gastro-entero-pancreatic neoplasms (GEP-NEN) derived from patients undergoing surgery for neuroendocrine neoplasia. This study will allow us to define the success rate in the generation of organoids from gastro-entero-pancreatic neoplasms (GEP-NEN).

SUMMARY:
Observational, prospective, feasibility pilot study of the preparation of organoids starting from tumor tissue and surrounding healthy tissue, collected during surgery, performed according to standard clinical practice.

DETAILED DESCRIPTION:
Given the need for the use of experimental models that mimic the tumor of origin

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age;
* diagnosis of GEP-NEN carried out via histological investigation or via positivity to the uptake PET-CT with 68Ga-peptides;
* availability of adequate material for the preparation of organoid cultures, derived from surgery;
* written informed consent.

Exclusion Criteria:

* previous chemotherapy treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients affected by GEP-NEN undergoing treatment will be enrolled in this study surgery to remove the tumor
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-11-03 (Estimated)

PRIMARY OUTCOMES:
Set up of at least 10 organoid cultures | 42 months
  The organoids will be generated from tumor tissue samples and surrounding healthy tissue obtained from patients affected by GEP-NEN (who meet the inclusion/exclusion criteria) collected, according to clinical practice, during tumor resection surgery. Only the excess material after carrying out all the investigations necessary for the correct diagnosis histological analysis can be used for the purpose of the project

CONTACTS AND LOCATIONS:
Overall Officials: Laura Monteonofrio, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy